CLINICAL TRIAL: NCT05231031
Title: Effect of Breathing and Relaxation Exercises on Serum Cortisol Levels in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hady Atef Labib, Lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DM and Cortisol
Record Dates: First submitted 2022-01-16; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus; Stress
MeSH Terms: conditions — Diabetes Mellitus | interventions — Exercise; Breathing Exercises; Relaxation Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise (Active Comparator): This group received continuous aerobic exercise only in the form of walking on a treadmill 3 sessions/week for 6 weeks
  Interventions: Behavioral: Aerobic exercise
- Aerobic, Breathing exercises , and relaxation training (Experimental): This group received continuous aerobic exercise only in the form of walking on a treadmill 3 sessions/week for 6 weeks in addition to breathing exercises and relaxation training for the same period
  Interventions: Behavioral: Aerobic exercise; Behavioral: breathing exercise; Behavioral: Relaxation training

INTERVENTIONS:
Behavioral: Aerobic exercise — continuous aerobic exercise on a treadmill
Behavioral: breathing exercise — continuous aerobic exercise plus breathing exercise (Mindfulness)
  Arms: Aerobic, Breathing exercises , and relaxation training
Behavioral: Relaxation training — continuous aerobic exercise plus relaxation training
  Arms: Aerobic, Breathing exercises , and relaxation training

SUMMARY:
Background: Diabetes is a fast-growing health problem in Egypt with a significant impact on morbidity, mortality, and health care resources. Aim of the study: To assess the effect of breathing and relaxation exercises on serum cortisol levels in type 2 diabetic patients. Subject and Methods: sixty, type 2 diabetic patients for more than 5 years were selected from the outpatient clinic of the Faculty of Physical Therapy, Cairo University. Their age ranged from 40 to 50 years. Serum cortisol and blood glucose tests were done before the start of the study and after 6 weeks. The patients were randomly assigned into two equal groups in number (30 patients for each group) performed 3 sessions/week for 6 weeks. Group A received aerobic exercise in the form of walking on a treadmill, breathing exercise, and mindfulness meditation, and group B received continuous aerobic exercise only in the form of walking on a treadmill. ( The exercise program included 45 minutes and consist of warming up phase of slow walking on the treadmill for 5 minutes, training phase 35 minutes, and cooling down for 5 minutes) .

DETAILED DESCRIPTION:
Diabetes is a metabolic disorder that requires ongoing medical care through multi-factor risk reduction strategies in addition to blood sugar control. Continuing education and support for diabetes self-management are essential to prevent acute complications and reduce the risk of long-term complications. There is a lot of evidence supporting a number of interventions to improve diabetes outcomes.

Diabetes mellitus (DM) is a chronic metabolic disorder characterized by persistent hyperglycemia. This may be due to insufficient insulin secretion, resistance to the peripheral effects of insulin, or both. The synergistic effect of chronic hyperglycemia and other metabolic abnormalities in diabetic patients can cause damage to various organ systems, leading to disabling and life-threatening health complications.

The global prevalence of type 2 diabetes has increased from 8.3% in 2013 to 9.3% in 2019. This increase has been higher in lower- to middle-income countries compared to high-income ones. Diabetes treatment includes behavioral and pharmacological approaches. Globally, it is estimated that only 23% (30% in Latin America) of people with diabetes have reached the set target. However, it is a challenge for treating physicians to choose a treatment that is tailored to each patient.

Egypt is the ninth-largest country in terms of type 2 diabetes mellitus (T2DM) patients, according to the International Diabetes Federation (IDF). T2DM patients have increased threefold in the last 20 years, with a current prevalence of 15.6 percent among people aged 20 to 79.

T2DM is a metabolic disorder that has both microvascular and macrovascular consequences. Controlling blood glucose levels is linked to a lower risk of microvascular consequences (retinopathy, nephropathy, and neuropathy) as well as macrovascular issues (lower incidence of heart attacks, strokes, and better blood flow to the legs).

The World Health Organisation (WHO) defines diabetes as a "metabolic disorder of multiple etiology characterized by chronic hyperglycemia with disturbance of carbohydrate, fat, and protein metabolism resulting from defects in insulin secretion, insulin action, or both. " The most prevalent form of diabetes is type 2, as an estimated 90% of diabetes patients are diagnosed with this form, and the majority of the remaining 10% of patients have type 1 diabetes (T1D), although there are other rare types. There is a range of effective treatments that reduce hyperglycemia in T2D patients, which mediate their effects by improving insulin secretion or decreasing peripheral tissue insulin resistance.

Diabetes is a chronic metabolic disease that can negatively affect the quality of life. Psychological stress and negative emotions have a two-way effect on diabetes control. Stress increases the risk and severity of diabetes by stimulating the hypothalamus-pituitary-adrenal gland (HPA) and sympathetic nerve axis and parasympathetic nerve withdrawal, leading to cortisol, epinephrine, norepinephrine, growth hormone, glucagon, catecholamines, Prolactin, leptin, and neuropeptide Y. Chronic activation of the HPA axis is related to poor control of complications such as diabetes and diabetic neuropathy. Elevated levels of inflammatory cytokines lead to insulin resistance in patients with type 2 diabetes. Chronic psychological stress can lead to an increased risk of insulin resistance, high blood pressure, and cardiovascular events.

Psychological stress has been linked to the development of type 2 diabetes. Meditation exercise can be viewed as a combination of mindfulness intervention and physical activity. This may partly explain why meditation exercises have a more positive effect on type 2 diabetes than other active and non-exercise exercises. A large number of studies have shown that meditation exercise is effective for blood sugar control in patients with type 2 diabetes.

Meditation interventions were shown to have a significant effect on changing cortisol levels assessed from blood samples.

Mindfulness meditation-based strategies are simple, easy to grasp and practice, and do not incur an additional cost. Meditation-based therapies may offer immediate positive benefits in such individuals.

Deep breathing has been shown to have a positive impact on various factors like stress, anxiety, and negative aﬀect in numerous studies.

Breathing exercises, also known as "diaphragmatic breathing" or "deep breathing", are defined as effective comprehensive training of the body and mind to deal with stress and physical and mental conditions. Diaphragm breathing involves the contraction of the diaphragm, the expansion of the abdomen, and the deepening of inhalation and exhalation, thereby reducing the respiratory rate and maximizing the amount of gas in the blood. The benefits of diaphragmatic breathing have been studied in conjunction with meditation.

Physical activity is a broad term that applies to any physical movement or activity that requires energy consumption by skeletal muscles. Aerobic exercise is a specific subcategory of physical activity. It is characterized by the rhythmic and continuous exercise of a large number of muscles, which mainly relies on the energy production process produced by oxygen metabolism. The main goal of aerobic exercise is to improve or maintain cardiorespiratory fitness, that is, the ability of the circulatory system and respiratory system to supply oxygen during continuous exercise

Exercise as a regular physical activity is found to be an efficient influencer that would switch back most of the known type 2 diabetes mellitus factors toward healthier positions. Exercise is proven to have clinical benefits, such as improved insulin sensitivity, reductions in glycosylated hemoglobin (A1C), and increased peak oxygen consumption (VO2peak) which are definitely preventive toward diabetes. Exercise improves blood glucose control in type 2 diabetes, reduces cardiovascular risk factors, and regulates body weight by reducing body fat percentage and enhancing lean mass.

Aerobic exercise consists of continuous, rhythmic movement of large muscle groups, such as in walking, jogging, and cycling. The most recent ADA guidelines state that individual sessions of aerobic activity should ideally last at least 30 minutes per day and be performed 3 to 7 days of the week. Moderate to vigorous (65%-90% of maximum heart and rate) aerobic exercise training improves VO2max cardiac output, which is associated with substantially reduced cardiovascular and overall mortality risk in patients with type 2 diabetes.

According to a study published in "Psycho-neuroendocrinology", there is a clear link between the stress hormone cortisol and high blood sugar levels in patients with type 2 diabetes mellitus (T2DM) The researchers explained that in healthy people, cortisol naturally fluctuates throughout the day. This natural fluctuation usually peaks in the morning and falls at night. However, patients with type 2 diabetes have lower levels of cortisol during the day and higher levels of glucose higher serum cortisol levels are a risk factor for future incidence of diabetes.

Cortisol is a glucocorticoid produced by activating the hypothalamic-pituitary-adrenal axis. It is called the "stress hormone" because it plays a major role in the body's response to stress. The activation of the HPA axis and the increase in cortisol secretion are important and adaptive parts of the human stress response, which can promote survival. However, when the stressor is activated for a long time, the HPA axis will become dysregulated, causing abnormal cortisol secretion and negatively affecting the body. Cortisol inhibits inflammation and allergic reactions, has an immunosuppressive effect, and also affects metabolic processes through gluconeogenesis (the release of amino acids from proteins in skeletal muscle and bone), glycogenolysis, and lipolysis

This study was conducted to investigate the effect of breathing and relaxation exercises on serum cortisol levels in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* • Sixty diabetic patients (29 women and 31 men), their age between 45 and 65 years .

  * They had type 2 diabetes mellitus for more than 5years.
  * Their HbA1c value from 6.5% to 7.5%.
  * Stress scores on the Perceived stress scale are >13 in the eligibility check assessment.
  * All patients are under full medical supervision.
  * Their physical activity level is less than 30 minutes of aerobic training in the week.
  * Their body mass index ranged from 25 to 34.9. (overweight and obesity class I).

Exclusion Criteria:

* • Any patient is known to have an unstable medical condition and sleeping disorder.

  * Indication of receiving treatments for depression and anxiety.
  * Musculoskeletal or neurological conditions that might interfere with the execution or the assessment of the exercise.
  * Cushing's disease (hypercortisolism) or Addison's disease (hypocortisolism).
  * Hepatic diseases and dyslipidemia.
  * Patients with renal and vascular diseases.
  * Severe hypertensive patients (higher than 200/120 mmHg).
  * Any acute or chronic inflammatory disorder.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Fating blood glucose | 6 weeks
  blood sampling for blood glucose after 9 hours fasting
Serum cortisol level | 6 weeks
  blood sampling for cortisol at 8 am

SECONDARY OUTCOMES:
The perceived stress score (PSS) | 6 weeks
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived

CONTACTS AND LOCATIONS:
Overall Officials: Hady Atef, PhD, Principal Investigator — Cairo University
Locations (1):
- Alkasr Alaini hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After approval can be shared
Supporting Information: Study Protocol
Time Frame: 12 months
Access Criteria: will upload it to the journal of publication